CLINICAL TRIAL: NCT00628160
Title: Effects on Survival of Terlipressin Administration in Cirrhotic Patients With Severe Sepsis or Septic Shock. A Randomized, Open Labelled Controlled Trial
Brief Title: Terlipressin in Septic Shock in Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Vicente Arroyo Perez, Senior Hepatologist Consultant, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-SS-JFDEZ-1; EUDRACAT-2005-000439-56; 2005-000439-56 (EudraCT Number)
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cirrhosis; Septic Shock
Keywords: Septic shock; Cirrhosis; Survival
MeSH Terms: conditions — Liver Cirrhosis; Shock, Septic; Fibrosis | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terlipressin group (Experimental): Terlipressin in continuous infusion plus alpha adrenergic drugs (noradrenaline and/or dopamine in continuous infusion)
  Interventions: Drug: Terlipressin
- Control group (Active Comparator): Alpha adrenergic drugs (noradrenaline and/or dopamine in continuous infusion)
  Interventions: Drug: alpha adrenergic drugs

INTERVENTIONS:
Drug: Terlipressin — Terlipressin 2-12 mg/24h intravenously in continuous infusion. Duration: until 24h after shock resolution.
  Other Names: Glypressin
  Arms: Terlipressin group
Drug: alpha adrenergic drugs — Dopamine (1-20 µg/Kg/min) and/or norepinephrine (0.05-4 µg/Kg/min) until shock resolution
  Other Names: Dopamine and/or norepinephrine
  Arms: Control group

SUMMARY:
Septic shock is a frequent and severe complication in cirrhosis. Current mortality rate ranges between 50 and 80% of cases. Refractory shock, hepatorenal failure and variceal bleeding are the main causes of death of these patients. Terlipressin administration could prevent these complications and improve survival in this setting.

Aim: To evaluate the effects of terlipressin administration on hospital survival in cirrhotic patients with severe sepsis or septic shock.

Methods: Prospective, open labelled, controlled trial evaluating 72 cirrhotic patients with severe sepsis or septic shock who will be randomized to receive terlipressin plus alpha-adrenergic drugs or only alpha-adrenergic drugs at shock diagnosis. Patients will be submitted to continuous systemic hemodynamic monitoring (S. Ganz catheter or Vigileo). Changes in vasoactive systems and cytokines levels will be also evaluated.

DETAILED DESCRIPTION:
Prospective, open labelled, RCT evaluating 72 cirrhotic patients with severe sepsis or septic shock (36 per arm) who were randomized to receive terlipressin plus alpha-adrenergic drugs or alpha-adrenergic drugs in the first 24h after septic shock diagnosis. Impact of terlipressin administration on shock reversal, changes in vasoactive systems, inflammatory response, incidence of variceal bleeding and type-1 HRS and ICU and hospital mortality was investigated

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years;
2. Diagnosis of cirrhosis based on histology or on clinical, laboratory and ultrasonographical data;
3. Diagnosis of septic shock based on the presence of data compatible with systemic inflammatory response syndrome, a mean arterial pressure below 60 mmHg during more than 1 hour despite adequate fluid resuscitation, and need for circulatory support with vasopressor drugs.

Exclusion Criteria:

1. More than 24 hours of evolution of the shock;
2. Cardiac index < 2,5 l/min;
3. History of HIV infection or clinically relevant pulmonary, renal or cardiac disease except for atrial fibrillation;
4. Pregnancy;
5. Advanced hepatocellular carcinoma (Milan criteria);
6. Previous history of transplantation;
7. Uncontrolled gastrointestinal bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hospital survival | Hospitalization

SECONDARY OUTCOMES:
Refractory shock | ICU admission
Variceal bleeding | ICU admission
Hepatorenal syndrome | Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Javier Fernandez, MD, Principal Investigator — Hospital Clinic of Barcelona; Vicente Arroyo, MD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
We are currently writing the manuscript